CLINICAL TRIAL: NCT06967753
Title: Switch to Dolutegravir Plus Lamivudine Dual-therapy in Transgender Women Living With HIV on Virologically Suppressive Antiretroviral Therapy (TRANS-SWITCH)
Acronym: TRANS-SWITCH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UBATEC (Other)
Collaborators: ViiV Healthcare (Industry); Hospital Fernandez (Other)
Responsible Party: Principal Investigator, Martin Jaume, Principal Investigator, Hospital Fernandez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIISA 14399
Record Dates: First submitted 2025-04-20; First posted 2025-05-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: HIV; HIV-1
Keywords: dual therapy; dolutegravir; antiretroviral treatment
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This will be a single-arm study (Experimental): Enrolled participants will be switched to a dual therapy strategy consisting of 50-mg DTG plus 300-mg 3TC tablet (as a single pill fixed dose combination) orally administered once daily with or without food. No dose reductions, modifications in dosage, or changes in the frequency of dosing will be allowed in this study.
  Interventions: Drug: Dolutegravir 50 MG plus lamivudine 300 MG； Dolutegravir/lamivudine (50 MG/300 MG)

INTERVENTIONS:
Drug: Dolutegravir 50 MG plus lamivudine 300 MG； Dolutegravir/lamivudine (50 MG/300 MG) — Enrolled participants will be switched to a dual therapy regimen consisting of 50-mg DTG plus 300-mg 3TC tablet (as a single pill fixed dose combination) orally administered once daily with or without food. No dose reductions, modifications in dosage, or changes in the frequency of dosing will be allowed in this study.

SUMMARY:
This single-arm, open label study is aimed to assess efficacy and safety of dolutegravir plus lamivudine as a switch strategy among TGW with HIV receiving suppresive antiretroviral therapy.

DETAILED DESCRIPTION:
This is a phase IV, 48-week, prospective, open-label, and single arm study. Study population will include 50 TGW living with HIV on suppressive ART. Eligible participants will be switched to a 2DR base of DTG + 3TC once daily and follow-up period will be 48 weeks.

The study timeline will consist of:

* a selection period of up to 30 days,
* a 48-week treatment period,
* and a 4-week post-treatment follow-up period.

The aim of the study will be to explore the effectiveness, safety, and acceptability of DTG + 3TC dual therapy among TGW living with HIV.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older at the time of signing the informed consent.
2. Self-identified as TGW.
3. Documented HIV-1 infection as per local standard: HIV-1 positive serology by at least two different serological tests (rapid test, ELISA, Western Blot) or a plasma HIV RNA viral ≥1,000 copies/mL.
4. ART-experienced participant on uninterrupted, stable, and suppressive triple ART for at least 3 months prior to screening, including: a) Acceptable stable ART regimens prior to Screening include 2 NRTIs plus i) INSTI ii) NNRTI or iii) Boosted PI. b) Any prior switch, defined as a change of a single drug or multiple drugs, must have occurred due to tolerability and/or safety concerns or access to medications, or convenience/simplification and must not have been done for suspected or established treatment failure. The following switches, if they are the only switches, would not be considered a change in regimen. a) A switch from a PI boosted with ritonavir (RTV) to the same PI boosted with cobicistat is allowed (and vice versa). b) A switch from 3TC to emtricitabine (FTC) (and vice versa). c) A switch from tenofovir disoproxil fumarate (TDF) to tenofovir alafenamide (TAF) (and vice versa).
5. Documented evidence of at least two HIV-1 RNA pVL <50 copies/mL in the last 12 months. HIV-1 RNA pVL corresponding to the screening visit may be accepted as second measurement.
6. Evidence of HIV-1 RNA pVL <50 copies/mL at screening visit.
7. Do not have history of previous virological failure and/or evidence of resistance to DTG or 3TC as per protocol definition.
8. Participants must be able to understand and comply with protocol.
9. Written informed consent provided.

Exclusion Criteria:

1. History or presence of hypersensitivity to any of the study drugs or their components.
2. Evidence of known acute or chronic viral hepatitis B (positive Hepatitis B surface antigen [HBsAg]) or hepatitis C (detectable plasma HCV RNA viral load). Participants with chronic Hepatitis B (positive HBsAg) or Hepatitis C (positive plasma HCV RNA viral load) will be excluded. Individuals with evidence of previous Hepatitis B (positive for Hepatitis B core antibody [HBcAc] but negative HBsAg may be included on the trial. Individuals with positive anti-HCV antibodies but with non-detectable plasma HCV RNA (previously treated or spontaneously cleared HCV) may be included in the study.
3. Evidence of untreated syphilis infection (positive VDRL at screening without clear documentation of treatment). Participants who are at least 7 days post completed treatment are eligible.
4. Evidence of an active centers for disease control and prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy. Historical or current CD4 cell counts less than 200 cells/millimeter are not exclusionary. Those individuals who are stable and receiving appropriate treatment for an HIV/AIDS-associated disease can be considered for the study.
5. Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected noninvasive cutaneous squamous cell carcinoma, or anal or penile intraepithelial neoplasia.
6. Participants with severe hepatic impairment (Class C) as determined by Child Pugh classification.
7. Any evidence of preexisting viral resistance based on the presence of any NRTI or INSTI major resistance associated mutation as per IAS-USA 2022 resistance panel in any historical resistance test result. 3TC resistance is considered in the presence of the M184V/I and/or K65R and/or Q151M mutations. DTG resistance is considered in the presence of the G118R, E138A/K/TG140A/C/R/S, Q148H/K/R, S153F/Y, N155H, or R263K mutations.
8. Participants who, as per the investigator's judgment, poses a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk.
9. Receiving other medications with relevant interactions with DTG and/or 3TC.
10. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of screening.
11. Treatment with any of the following agents within 28 days of screening: radiation therapy, cytotoxic chemotherapeutic agents, any systemic immune suppressant.
12. Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of the study drug.
13. Laboratory tests performed at the screening visit show any of the following results: a. Any verified Grade 4 laboratory abnormality. b. Hemoglobin <9.0 g/dL c. Absolute neutrophil count <750 cel/µL d. Platelet count <80,000 cel/mm3 e. Creatinine clearance <30 mL/min according to the Cockroft-Gault formula. f. Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN) or ALT ≥3 times ULN and bilirubin ≥1.5 times ULN (with >35% direct bilirubin).
14. Any condition (including but not limited to the abuse of alcohol or drugs) which in the opinion of the investigator could compromise the participant's safety or adherence to the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender Women
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Virological efficacy | 48 weeks
  Proportion of participants with HIV-1 RNA pVL >= 50 copies/mL at 48 weeks of treatment as per the intent-to-treat exposed (ITT-E) snapshot FDA algorithm.

SECONDARY OUTCOMES:
Virological efficacy | 48 weeks
  Proportion of participants with HIV-1 RNA pVL >= 50 copies/mL at week 48 as per-protocol (PP) analysis.
Virological efficacy | 24 weeks
  Proportion of participants with HIV-1 RNA pVL >= 50 copies/mL at 24 weeks of treatment as per the ITT-E snapshot FDA algorithm.
Changes in CD4+ count | 24 and 48 weeks
  Absolute values and change from baseline in CD4+ lymphocyte count at weeks 24 and 48.
Safety - Adverse Events (including Serious Adverse Events and Adverse Events Leading to Discontinuation) | 48 weeks
  Number of participants with any AEs, SAEs, AEs by their severity grades, and AEs leading to discontinuation through 48 weeks. AE will be evaluated by the investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death).
Changes in lipid profile measurements | 24 and 48 weeks
  Change from baseline in serum or plasma total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol and triglycerides at weeks 24 and 48. Fasting blood samples will be collected to assess total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides. Baseline value is defined as the latest pre-dose assessment. Change from baseline is defined as post-dose visit value minus baseline value.
Changes in Kidney Function measurements | 24 and 48 weeks
  Change from baseline in plasma creatinine at weeks 24 and 48. Blood samples will be collected to perform assess serum or plasma creatinine at week 24 and 48. Baseline value is defined as the latest pre-dose assessment. Change from baseline was calculated as post-dose visit value minus baseline value.
Changes in Body Weight | 24 and 48 weeks
  Change from baseline in absolute body weight and Body Mass Index (BMI) at weeks 24 and 48. Baseline value is defined as the latest pre-dose assessment.
Changes in Bone Mineral Density | 48 weeks
  Percent change from baseline in Bone Mineral Density (BMD) of the hip and lumber spine to week 48. BMD will be evaluated by dual-energy x-ray absorptiometry (DEXA) scans at study baseline and week 48.
Emerging resistance to study drugs | 48 weeks
  Number of participants with confirmed virological failure as per the protocol with observed genotypic resistance to DTG and/or 3TC.
Quality of LIfe | Weeks 4, 24 and 48
  Change from Baseline in health-related quality of life using European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) and Patient Health Questionnaire-9 (PHQ-9) at baseline and weeks 4, 24 and 48.
Treatment acceptance | Weeks 4, 24 and 48
  Change from Baseline in HIV treatment acceptance using Treatment Satisfaction Questionnaire change version (HIVTSQc) and Chronic Treatment Acceptance questionnaire (ACCEPT) at baseline and weeks 4, 24 and 48.
Treatment Adherence | Weeks 4, 12, 24, 36 and 48.
  Adherence using the ACTG adherence questionnaire at baseline and weeks 4, 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Martín Jaume, MD, Principal Investigator — Hospital Fernández, Infectious Diseases Division
Locations (1):
- Hospital General de Agudos Dr. Juan A. Fernández, Infectious Diseases Division, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided